CLINICAL TRIAL: NCT01353196
Title: Asymptomatic Carotid Stenosis: Cognitive Function and Plaque Correlates
Acronym: ACCOF
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CARA-024-10S
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Cognitive Manifestations
Keywords: carotid; atherosclerosis; cognitive function
MeSH Terms: conditions — Neurobehavioral Manifestations; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples for inflammatory markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- stenosis: carotid stenosis
- no stenosis: no stenosis

SUMMARY:
Carotid artery plaques are known to cause stroke. Cognitive impairment is an insidious but poorly understood problem in patients with carotid plaques. Cognitive function describes how people perform mental processes such as thinking, learning and problem solving. Asymptomatic carotid plaques may affect 1 million Veterans who may be at risk for cognitive impairment. In this study, the investigators will uncover the extent of cognitive impairment in Veterans with carotid stenosis who are currently labeled "asymptomatic". Programs to prevent or mitigate cognitive impairment will depend on identifying the mechanisms by which this occurs. The investigators will use sophisticated 3D imaging techniques developed by the group to measure the structure and composition of plaques, number of particles breaking off from them, blood levels of chemicals that could disrupt them, and blood flow restriction to the brain from them. This will help identify patients at risk for cognitive impairment who may benefit from preventative measures and improve selection of patients to decrease unnecessary surgical procedures.

DETAILED DESCRIPTION:
Carotid artery stenosis is a well-known cause of atheroembolic stroke. Stroke prevention in these patients has been the focus of intense investigation. Cognitive impairment is a more insidious but poorly understood outcome in patients with "asymptomatic" carotid stenosis who have not suffered a stroke. Cognitive function describes how a person produces and controls mental processes such as thinking, learning, and problem solving. It is an important outcome measure that affects patient well-being and their ability to live independent productive lies. It is well-known that cognitive impairment coexists in patients with stroke from carotid stenosis. However, isolated cognitive deficits in patients with asymptomatic carotid stenosis have not been looked for, and have therefore not been reported in any detail. Asymptomatic carotid stenosis affects 2-12% of people. With 23.4 million Veterans in the country, at least 1 million (4.3%) have asymptomatic carotid stenosis and are at risk for cognitive impairment. A subset analysis of the Cardiovascular Health Study found cognitive decline in 34% of 32 patients with asymptomatic carotid stenosis. In this proposal, the investigators will define the extent of initial and progressive cognitive impairment in Veterans with carotid stenosis who are currently labeled as "asymptomatic" in the absence of a focal neurologic deficit (stroke, transient ischemic attack). Programs to prevent, postpone, or mitigate cognitive impairment in patients with carotid stenosis will depend on the identification of mediators for cognitive impairment. Microembolic brain injury and cerebral hypoperfusion have been associated with cognitive impairment in elderly individuals.

Therefore plaque architecture, plaque composition, microembolic counts, serum inflammatory markers, and cerebral hypoperfusion are likely mediators of impaired cognition in patients with asymptomatic carotid stenosis. As part of this proposal, the investigators will identify the biological mechanisms by which carotid stenosis could result in cognitive impairment.

The goal of this proposal is to perform a systematic, adequately powered study to measure the magnitude of cognitive impairment in asymptomatic carotid stenosis, its impact on quality of life, and its potential pathophysiological mechanisms. Information from this study will define an unsuspected morbidity of carotid stenosis and identify subsets of patients at risk for cognitive impairment. It will form the foundation for future studies on prevention, pre-emptive treatment, or rehabilitation of patients with carotid stenosis. It will also improve the selection of patients with carotid stenosis to decrease unnecessary revascularization procedures.

Specific Aim 1 will assess if patients with asymptomatic carotid stenosis differ in cognitive function compared to age-matched controls without carotid stenosis but with similar vascular risk profiles. The investigators hypothesize that in patients with asymptomatic carotid stenosis 50% who survive stroke free for 2 years; the change in overall and domain-specific cognitive function will be significantly different compared to those without stenosis. The study will recruit 284 subjects and will detect a clinically significant difference in cognitive score with 90% power. The investigators will use a novel battery of cognitive tests specifically developed to address the unique issues relating to carotid stenosis.

Specific Aim 2 will define plaque-morphometric, biologic, and hemodynamic characteristics that correlate with cognitive impairment in patients with asymptomatic carotid stenosis. The investigators hypothesize that carotid plaque architecture, plaque composition, microembolic counts, serum pro-inflammatory markers, and cerebral hypoperfusion could each mediate cognitive decline over a 2-year follow-up period. The investigators will implement a novel clinical 3D B-mode ultrasound imaging technique developed to obtain reliable serial plaque measurements.

Specific Aim 3 will measure the impact of cognitive impairment on quality of life. The investigators hypothesize that at 2 years, regardless of plaque features, cognitive impairment will correlate with a reduction in health-related quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic 50% carotid stenosis or more

Exclusion Criteria:

* previous stroke or transient ischemic attack (TIA)
* severe medical illness that would interfere with evaluation of outcomes or reduce the likelihood of a 2-year follow-up
* carotid occlusion
* patients scheduled for carotid revascularization procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for the study will have asymptomatic >=50% carotid stenosis
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-05-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brajesh K Lal, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lal BK, Dux MC, Sikdar S, Goldstein C, Khan AA, Yokemick J, Zhao L. Asymptomatic carotid stenosis is associated with cognitive impairment. J Vasc Surg. 2017 Oct;66(4):1083-1092. doi: 10.1016/j.jvs.2017.04.038. Epub 2017 Jul 14. PMID 28712815

RESULTS

PARTICIPANT FLOW:
Groups:
- Stenosis: participants with carotid stenosis
- no Stenosis: participants with no carotid artery stenosis
Period: Overall Study
Arm/Group | Stenosis | no Stenosis
Started | 100 | 70
Completed | 71 | 59
Not Completed | 29 | 11

BASELINE CHARACTERISTICS:
Groups:
- no Stenosis: no carotid artery stenosis
- Total: Total of all reporting groups
Arm/Group | Stenosis | no Stenosis | Total
Number analyzed (Participants) | 100 | 70 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 74 | 44 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10) | 50 (10) | 50 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 99 | 68 | 167
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 34 | 58
  White | 76 | 36 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Composite cognitive function [Mean (Standard Deviation); unit: units on a scale] — 0 = worst 100 = best
  units on a scale | 45.5 (6.0) | 47.9 (5.0) | 46.0 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Composite Cognitive Score
Description: composite of multiple cognitive function test scores scores are reported as mean +/- standard deviation 0 = worst 100 = best
Time Frame: 2 years
Population: Participants that did not complete the study or missing key data elements were excluded from the overall analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenosis | no Stenosis
Number analyzed (Participants) | 82 | 62
units on a scale | 45.5 (6.0) | 47.9 (5.0)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Stenosis | no Stenosis
All-Cause Mortality (participants affected / at risk) | 18/100 | 11/70
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/70
Other Adverse Events (participants affected / at risk) | 0/100 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT01353196/Prot_SAP_000.pdf